CLINICAL TRIAL: NCT07312890
Title: Bedside Observation by Clinical Ultrasound for Stomach Expansion
Acronym: BOCUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Saint Joseph Saint Luc de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BOCUSE
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Enteral Feeding Intolerance
Keywords: Enteral feeding intolerance; Gastric antral area

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monitoring of enteral nutrition intolerance (Other): Monitoring of enteral nutrition intolerance : presence of regurgitation or vomiting, and interruption or reduction of enteral nutrition flow rates over a 7-day period. Gastric ultrasound with measurement of the antral area
  Interventions: Other: Gastric ultrasound with measurement of the antral area

INTERVENTIONS:
Other: Gastric ultrasound with measurement of the antral area — Gastric ultrasound with measurement of the antral area

SUMMARY:
The objective of the BOCUSE study is to demonstrate a relationship between an early ultrasound measurement of the gastric antral area and the subsequent occurrence of poor gastric tolerance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Predicted mechanical ventilation ≥ 48 hours
* Initiation of enteral nutrition via nasogastric or orogastric tube for ≥ 48 hours
* Free and informed consent obtained from the patient's relative or legal representative, or inclusion in an emergency situation

Exclusion Criteria:

* History of major gastric surgery (bypass, total gastrectomy, biliopancreatic diversion)
* Enteral nutrition via nasogastric or orogastric tube > 96 hours
* Initiation of enteral nutrition before intubation
* Feeding via gastrostomy, jejunostomy, or jejunal tube
* Pregnancy
* Prognosis considered terminal
* No ultrasound window available
* Legally protected adults (under curatorship, guardianship, or judicial protection)
* No social security coverage
* Patient under State Medical Aid (AME)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-25 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-01-25 (Estimated)

PRIMARY OUTCOMES:
Enteral nutrition intolerance | Within 7 days following the gastric ultrasound
  Presence of regurgitation and/or vomiting and/or interruption or reduction of enteral nutrition flow rates

SECONDARY OUTCOMES:
Occurrence of VAP | From H0 until ICU discharge, up to 3 months
  Occurrence of Ventilator Associated Pneumonia
Mortality | At ICU discharge, at 28 days, and at 3 months
  Mortality at ICU discharge, at day 28, and at 3 months
Duration of mechanical ventilation | From H0 until ICU discharge, up to 3 months
  Number of days on mechanical ventilation
Number of ventilator-free days | Day 28, 3 months
  Number of ventilator-free days at day 28 and 3 months
Length of stay in the ICU | From ICU admission until ICU discharge, up to 3 months
  Length of ICU stay (in days)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Saint Joseph Saint Luc, Lyon, France

IPD SHARING:
Plan to Share IPD: No